CLINICAL TRIAL: NCT05295888
Title: Evaluation of Temporal Interference in Target Engagement of Subgenual Cingulate Cortex in the Treatment of Major Depressive Disorder
Brief Title: Temporal Interference and Depression
Acronym: TI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Northeastern University (Other); Centre for Addiction and Mental Health (Other); Charite University, Berlin, Germany (Other); Toronto Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-152
Record Dates: First submitted 2021-10-08; First posted 2022-03-25 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: This is a pilot, sham-controlled, quadruple-blind clinical trial to demonstrate target engagement of SCC with TI, as well as assess feasibility, safety, tolerability, and preliminary therapeutic efficacy of TI stimulation in patients with MDD.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The following roles will be blinded: i) Investigators and care providers; ii) Enrolled participants; iii) Outcome assessors; iv) MRI technician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): 130Hz TI stimulation (total 30 min) + mood induction paradigm: ramp-up (30 sec) => stimulation (130Hz, 2mA per electrode pair, 4mA total, 29 min) => ramp-down (30 sec)
  Interventions: Device: Temporal Interference stimulation
- Sham Arm (Sham Comparator): Sham stimulation (total 30 min) + mood induction paradigm: ramp-up (30 sec) => ramp-down (30 sec) => stimulation (130Hz, 0mA, 29 min)
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Temporal Interference stimulation — TI involves simultaneous delivery of independent currents to the brain at slightly different kHz frequencies, which are individually too high to recruit neural firing. However, the difference ('beat') frequency where the currents overlap (i.e., temporally interfered) is low enough to drive neural activity. The interferometrically derived low frequencies have been demonstrated to activate neurons at a selected focus without activation of surrounding regions in awake mice. The safety of the TI paradigm has been demonstrated in over 60 healthy human volunteers, and finite element modeling of simulations of TI fields in human anatomical models suggests that large subcortical structures such as the hippocampus or SCC could be selectively targeted. However, the precise TI parameters for selective engagement of SCC in healthy participants and in MDD is currently unknown.
  Arms: Experimental Arm
Device: Sham stimulation — Electrodes will be placed in the same location on the head as that for the TI intervention; 0 mA of electrical current will be delivered to the brain (compared to 2 mA in the active intervention arm), therefore it is expected to elicit no changes in neural activity.
  Arms: Sham Arm

SUMMARY:
Major Depressive Disorder (MDD) has a high prevalence, is the leading cause of disability, and currently available interventions are associated with side effects and high treatment resistance. There is an urgent need for the development of novel interventions for MDD with alternate mechanisms of action. Temporal Interference (TI) stimulation is a newly emerging form of transcranial alternating current stimulation (tACS) that involves the application of two high-frequency currents at slightly different kHz frequencies. Since neurons, due to their intrinsic low-pass filtering, do not respond to high frequencies (i.e. > 100 Hz), TI relies on the 'beat' interaction leading to neuromodulation at any given location, resulting in a much smaller focus and allowing for better targeting. The subgenual cingulate cortex (SCC) appears to be critical in the pathophysiology of depression and treatment response, especially in treatment-resistant cases. Non-invasive treatments, however, are not able to accurately target SCC due to its deep location within the brain. In this trial, 30 participants meeting the diagnostic criteria for MDD will be randomized to receive 10 sessions of 130 Hz TI delivered daily for 30 minutes, or 10 sessions of sham stimulation. During the stimulation, participants will be watching emotional film clips to enhance target engagement. The investigators will collect metrics of SCC target engagement using the resting-state fMRI and EEG technologies, and determine feasibility, tolerability, safety, and therapeutic efficacy of TI stimulation in MDD. The results of this trial will inform the TI technology as a therapeutic tool for network-based psychiatric disorders, including MDD, and be vital for the design and development of a large-scale randomized-controlled trial.

ELIGIBILITY:
Inclusion Criteria - Patients will be included if they:

1. provide written informed consent before initiation of any study-related procedures
2. are outpatients
3. meet the DSM-5 criteria for major depressive disorder (MDD) with a current major depressive episode (MDE) without psychotic features as confirmed at Screening by the Mini International Neuropsychiatric Interview (MINI)
4. are male or female, 18 to 65 years of age (inclusive) at screening
5. have a Montgomery-Åsberg Depression Rating Scale (MADRS) total score of ≥ 20 (moderate to severe depression) at screening
6. have had no increase or initiation of any psychotropic medication in the 4 weeks prior to screening
7. able to adhere to the treatment schedule
8. pass the TI adult safety screening questionnaire
9. are able to understand and comply with the requirements of the study, as judged by the investigator(s)

Exclusion Criteria - Patients will be excluded if they:

1. have an acute alcohol or substance use disorder, withdrawal symptoms requiring detoxification, or went through detoxification treatment (inpatient or outpatient) within 3 months before Screening, as obtained from MINI, Module I (Alcohol Use Disorder) and Module J (Substance Use Disorder, Non-Alcohol) assessed at Screening
2. have a concomitant major unstable medical illness, active hepatitis B virus (HBV), hepatitis C virus (HPC), human immunodeficiency virus (HIV), active COVID-19 infection, cardiac pacemaker or implanted medication pump, as per medical history provided by the participant
3. have active suicidal intent, confirmed by a 'Yes' response to Question B3 AND either Question B10 or B11, obtained from the MINI Suicidality, Module B (Suicidality), OR confirmed by the MADRS item #10 score ≥ 4, both assessed at Screening
4. have a current clinical diagnosis of autism, dementia, or intellectual disability
5. take medications prohibited by the protocol. Medications will be reviewed by the responsible MD
6. are pregnant or lactating
7. have any prior or current diagnosis of bipolar I or II disorder, MDD with psychotic features, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms as obtained from MINI, Module C (Manic and Hypomanic Episodes) and Module K (Psychotic Disorders and Mood Disorders with Psychotic Features) assessed at Screening
8. have any prior or current diagnosis of obsessive-compulsive disorder, post-traumatic stress disorder (current or within the last year), confirmed by MINI and assessed by a study investigator to be primary and causing greater impairment than MDD
9. have a diagnosis of any personality disorder, and assessed by a study investigator to be primary and causing greater impairment than MDD
10. have received TI for any previous indication due to the potential compromise of subject blinding
11. have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space-occupying brain lesion, any history of seizure except those therapeutically induced by ECT or a febrile seizure of infancy, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than 5 minutes, current history of poorly controlled migraines including chronic medication for migraine prevention
12. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
13. if participating in psychotherapy, have NOT been in stable treatment for at least 3 months prior to entry into the study or anticipate change in the frequency of therapeutic sessions or therapeutic focus over the duration of the study
14. have a clinically significant laboratory abnormality, in the opinion of one of the principal investigators or study physicians
15. currently take medications that potentially limit the TI efficacy
16. have a non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with an interview)
17. have a clinical finding that is unstable or that, in the opinion of the investigator(s), would be negatively affected by the study medication or that would affect the study medication (e.g., diabetes mellitus, hypertension, unstable angina)
18. have uncorrected hypothyroidism or hyperthyroidism. Subjects needing a thyroid hormone supplement to treat hypothyroidism will be excluded if they have NOT been on a stable dose of the medication for 30 days prior to enrolment
19. have any other condition that, in the opinion of the investigator(s), would adversely affect the subject's ability to complete the study or its measure
20. wear a hairstyle or headdress at the time of the stimulation that prevents electrode contact with the scalp or would interfere with the stimulation (e.g., thick or curly hair)
21. have any contraindications for receiving TI or undergoing MRI scans (e.g., hip circumference >180 cm or metal in the body)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Neuroimaging - Signal variance | End of 2nd week of intervention
  Signal variance within SCC to demonstrate SCC target engagement to TI stimulation
Neuroimaging - Functional connectivity | End of 2nd week of intervention
  Seed-based resting-state functional connectivity of SCC to demonstrate SCC target engagement to TI stimulation
Neuroimaging - Anatomical connectivity | End of 2nd week of intervention
  Anatomical connectivity of SCC to demonstrate SCC target engagement to TI stimulation
Neuroimaging - Perfusion metrics | End of 2nd week of intervention
  Cerebral blood flow within SCC to demonstrate SCC target engagement to TI stimulation

SECONDARY OUTCOMES:
Clinical change in depression symptoms | Baseline, end of 1st week of intervention, end of 2nd week of intervention, 1 week post-intervention, and 4 weeks post-intervention
  Change in symptoms of depression measured by the 17-item Hamilton Depression Rating Scale (HAM-D); scores range from 0 to 53, and higher scores indicate more severe depression symptoms.
Clinical change in depression symptoms | Baseline, each intervention visit (5 times/week for 2 weeks), 1 week post-intervention, and 4 weeks post-intervention
  Change in symptoms of depression measured by the 16-item Quick Inventory of Depressive Symptomatology; scores range from 0 to 48, and higher scores indicate more severe depression symptoms.
EEG Signals - Time domain features | Baseline, end of 1st week of intervention, and end of 2nd week of intervention
  Changes in time domain features of gamma oscillation on resting-state EEG Changes in time domain features of theta oscillation on resting-state EEG
EEG Signals - Frequency domain features | Baseline, end of 1st week of intervention, and end of 2nd week of intervention
  Changes in frequency domain features of gamma oscillation on resting-state EEG Changes in frequency domain features of theta oscillation on resting-state EEG
EEG Signals - Functional connectivity | Baseline, end of 1st week of intervention, and end of 2nd week of intervention
  Changes in functional connectivity on resting-state EEG
Correlation between EEG and depression symptoms | Baseline, end of 1st week of intervention, and end of 2nd week of intervention
  Correlation between changes in features of gamma or theta oscillations (EEG) and changes in depression symptoms measured by the HAM-D
EEG Signals - MMN event-related potential | Baseline, end of 1st week of intervention, and end of 2nd week of intervention
  Changes in mismatch negativity (MMN) event-related potential amplitude and latency
Tolerability - Adverse events | End of 1st week of intervention, end of 2nd week of intervention, 1 week post-intervention, and 4 weeks post-intervention
  Incidence of treatment-emergent adverse events
Trial Feasibility - Dropout rate | End of 1st week of intervention, end of 2nd week of intervention, 1 week post-intervention, and 4 weeks post-intervention
  The proportion of participants who discontinue participation in the study before completion
Trial Feasibility - Recruitment rate | Enrollment
  The number of participants enrolled into the study per month
Trial Feasibility - Intervention adherence | End of 2nd week of intervention
  Percentage of participants who completed ≥80% of scheduled intervention sessions

CONTACTS AND LOCATIONS:
Overall Officials: Venkat Bhat, MD MSc, Principal Investigator — Unity Health Toronto
Locations (1):
- Interventional Psychiatry Program, St. Michael's Hospital - Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demchenko I, Rampersad S, Datta A, Horn A, Churchill NW, Kennedy SH, Krishnan S, Rueda A, Schweizer TA, Griffiths JD, Boyden ES, Santarnecchi E, Bhat V. Target engagement of the subgenual anterior cingulate cortex with transcranial temporal interference stimulation in major depressive disorder: a protocol for a randomized sham-controlled trial. Front Neurosci. 2024 Aug 29;18:1390250. doi: 10.3389/fnins.2024.1390250. eCollection 2024. PMID 39268031